CLINICAL TRIAL: NCT03305549
Title: Recovery After Dialysis-Requiring Acute Kidney Injury Pilot Study
Brief Title: Recovery After Dialysis-Requiring Acute Kidney Injury
Acronym: RAD-AKI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study stopped because sufficient pilot data collected to proceed to next clinical trial.
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F32DK115030 (NIH); F32DK115030 (NIH)
Record Dates: First submitted 2017-09-29; First posted 2017-10-10 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Acute Kidney Injury
Keywords: Dialysis-requiring Acute Kidney Injury; Renal Recovery
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Intervention Model Description: Pilot 2-arm parallel-comparison randomized clinical trial comparing TIW dialysis (control) to a "conservative dialysis strategy."
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TIW Dialysis Strategy (Active Comparator): Conventional thrice-weekly acute intermittent hemodialysis treatment schedule.
  Interventions: Other: TIW dialysis strategy
- Conservative Dialysis Strategy (Experimental): Conservative acute intermittent hemodialysis strategy, in which hemodialysis is not continued unless specific metabolic or clinical indications for RRT are present.
  Interventions: Other: Conservative dialysis strategy

INTERVENTIONS:
Other: Conservative dialysis strategy — Participants will receive RRT only when meeting 1 of the following indications (patterned after the AKIKI trial's delayed RRT initiation arm):
  * Blood urea nitrogen >112 mg/dL (40 mmol/L)
  * Serum potassium concentration >6 mmol/L
  * Serum potassium concentration >5.5 mmol/L despite medical treatment (e.g., bicarbonate, glucose-insulin infusion, albuterol, diuretics, sodium polystyrene sulfonate)
  * Arterial blood gas pH <7.15 in a context of pure metabolic acidosis (PaCO2 <35 mmHg) or in a context of mixed acidosis with PaCO2 50 mmHg despite medical treatment to reverse respiratory acidosis (e.g., naloxone), or in the absence of an available arterial blood gas, serum bicarbonate <12 mmol/L
  * Acute pulmonary edema due to fluid overload, responsible for hypoxemia requiring oxygen flow rate >5 L/min to maintain SpO2 >95% or requiring FiO2 >50% in patients already on invasive or non-invasive mechanical ventilation and despite diuretic therapy
  Arms: Conservative Dialysis Strategy
Other: TIW dialysis strategy — Thrice-weekly acute intermittent hemodialysis schedule.
  Arms: TIW Dialysis Strategy

SUMMARY:
The Recovery After Dialysis-Requiring Acute Kidney Injury (RAD-AKI) Pilot Study is a 2-arm randomized clinical trial of hospitalized patients with dialysis-requiring acute kidney injury (RAD-AKI), comparing conventional thrice-weekly intermittent hemodialysis dialysis (control) to a "conservative dialysis strategy" in which hemodialysis is not continued unless specific metabolic or clinical indications for RRT are present. The overall hypothesis is that the current practice of thrice-weekly acute intermittent hemodialysis for AKI-D masks evidence of renal recovery and may actually delay or preclude recovery. The primary objective of this pilot study is to assess the safety and feasibility of the proposed intervention and study design.

DETAILED DESCRIPTION:
The recent landmark Artificial Kidney Initiation in Kidney Injury (AKIKI) trial showed that a delayed strategy for RRT initiation among patients with incident stage 3 AKI - in which RRT was delayed unless specific metabolic or clinical indications for RRT were present - was safe and averted the need for RRT in nearly half of the critically ill participants, in comparison to an early RRT initiation strategy. The hypothesis for this study is: for prevalent patients with established AKI-D, a conservative dialysis strategy - in which hemodialysis is not continued unless specific metabolic or clinical indications for RRT are present - will shorten time to RRT-independence and improve the likelihood of renal recovery.

The RAD-AKI Pilot Study is a 2-arm randomized clinical trial of hospitalized patients with dialysis-requiring acute kidney injury (RAD-AKI) that will compare conventional thrice-weekly intermittent hemodialysis dialysis (control) to a "conservative dialysis strategy." The primary objective of this pilot study is to assess the safety and feasibility of the proposed intervention and study design.

ELIGIBILITY:
Inclusion Criteria:

* Adult inpatients with AKI-D due to acute tubular necrosis who have already initiated renal replacement therapy
* If initiated on CRRT, patients will be eligible only if they have already tolerated 1 intermittent hemodialysis (IHD) session at the research site.
* If transferred from an outside hospital, eligible patients must have tolerated 1 IHD session at the research site prior to enrollment.
* Not requiring vasopressor support
* Not intubated and not having a supplemental oxygen requirement of >5 L/min via nasal cannula
* Treating MDs (nephrology and primary team attendings) and patient (or legally authorized representative) consent to enrollment

Exclusion Criteria:

* Diagnosis of end-stage renal disease (ESRD) or chronic dialysis prior to hospitalization
* Baseline estimated glomerular filtration rate (eGFR) <15 mL/min/1.73m2
* Liver transplant unit patients
* Patients who underwent kidney transplantation during index hospitalization
* Cause of AKI-D is complete nephrectomy
* Current pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2019-11-13 (Actual)

PRIMARY OUTCOMES:
Protocol adherence [feasibility measure] | Through completion of active study participation (anticipated <2 weeks for each participant)
  Number of times a participant in the "conservative dialysis" arm receives dialysis despite not meeting one of the pre-specified indications for dialysis, number of times a participant in the "TIW dialysis" arm is dialyzed off-schedule
Number of participants with adverse events in each arm [safety measure] | Through completion of active study participation (anticipated <2 weeks for each participant)
  Both serious and non-serious adverse events will be monitored, including arrhythmias due to metabolic disturbances, death, emergent dialysis needs, and transfer to ICU or intubation after enrollment

SECONDARY OUTCOMES:
Patient-reported symptoms | Through completion of active study participation (anticipated <2 weeks for each participant)
  Survey will assess dyspnea, light-headedness, intradialytic cramping, pain and impaired mobility due to edema
Hospital length of stay | Through completion of active study participation (anticipated <2 weeks for each participant)
  Length of inpatient admission, starting after study enrollment
Recovery status at 30, 60, and 90 days after dialysis initiation | From enrollment to 90 days after dialysis initiation for each patient
  Assessment of recovery status via phone call or e-mail contact
Screen-to-enroll ratio [feasibility measure] | Through study completion (anticipated 2 years total)
  Ratio of number of participants who meet eligibility criteria to number of participants who actually enroll into the study

CONTACTS AND LOCATIONS:
Overall Officials: Chi-yuan Hsu, MD, MSc, Principal Investigator — University of California, San Francisco; Kathleen Liu, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Medical Center Moffitt-Long Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No